CLINICAL TRIAL: NCT03887338
Title: Systematic Laryngoscopic Evaluation of Upper Airways in Ventilated Amyotrophic Lateral Sclerosis (ALS) Patients in Portugal and in Norway
Brief Title: Systematic Laryngoscopic Evaluation of Upper Airways in Ventilated ALS Patients in Portugal and in Norway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tiina Maarit Andersen (Other)
Collaborators: University of Trás-os-Montes and Alto Douro (Other); Universidade do Porto (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor-Investigator, Tiina Maarit Andersen, Respiratory Physiotherapist, PhD, Haukeland University Hospital
Organization: Haukeland University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/1306; 39/2016 (Other: Centro Hospitalar Trás-os-Montes e Alto Douro, Vila Real)
Record Dates: First submitted 2019-03-15; First posted 2019-03-22 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Noninvasive Ventilation; Laryngoscopy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: All the subjects will receive the same intervention, and they will be examined both prior to the intervention, one month after and three months after the intervention. They will act as they own controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIV settings titration (Other): Transnasal Fiberoptic Laryngoscopy will be used during ongoing NIV setting titration. Aim is to titrate NIV setting to be more optimal for laryngeal responses.
  Interventions: Other: Transnasal Fiberoptic Laryngoscopy

INTERVENTIONS:
Other: Transnasal Fiberoptic Laryngoscopy — Use of Transnasal Fiberoptic Laryngoscopy during NIV titration to optimalize the NIV settings to laryngeal responses during the NIV treatment.

SUMMARY:
The study examines if titration of Non-Invasive mechanical ventilation (NIV) settings during ongoing laryngoscopic visualization can improve the compliance of NIV in subjects with Amyotrophic Lateral Sclerosis (ALS). The study is a multicentre study between Norwegian National Advisory Unit on Long-term Mechanical Ventilation at the Thoracic Department, Haukeland University Hospital, Bergen, Norway and Centro Hospital Tras-os-Montes e Alto Douro, Vila Real, Portugal.

DETAILED DESCRIPTION:
ALS, amyotrophic lateral sclerosis, is a rare and fatal disease causing gradual loss of motor neurons and thus loss of function in all skeletal muscle, eventually also in the breathing muscles, leading to respiratory failure and ultimately death. There is no causal treatment. The treatment provided aims to improve life quality as long as possible. Non-invasive ventilation (NIV) compensates for respiratory failure as breathing deteriorates.

ALS patients with bulbar innervated muscle dysfunction (mouth, tongue, jaw, throat, larynx) have poor compliance to the use of NIV. It is not completely understood why bulbar ALS patients fails NIV, although the upper airways have been a suggested cause also of this treatment failure. The investigators in the Norwegian study group has previously examined laryngeal response patterns (using transnasal fiberoptic laryngoscopy ) during mechanically assisted cough in ALS. The studies revealed that Transnasal fiberoptic laryngoscopy was safely performed with ongoing mechanically assisted cough, and it appeared a feasible tool to visualize the laryngeal responses to mechanical cough therapy.

The further hypothesis is that the use of transnasal fiberoptic laryngoscopy during ongoing NIV titration could improve the compliance of NIV treatment in ALS.

Since ALS is a relatively rare disease and it is difficult to perform large clinical studies, a project group has been established and agreed to a common protocol of a population-based multicenter-study including two hospitals, in Bergen in Norway and Vila Real in Portugal.

Aims of the study are:

To investigate the feasibility of video-recorded Transnasal fiberoptic laryngoscopic evaluation of the upper airways applied during NIV titration, and to describe the upper airway responses to NIV treatment in patients with ALS.

To explore whether the endoscopic view of the upper airways will influence the titration of NIV settings in ALS patients.

To explore whether NIV titration with endoscopic evaluation will influence NIV compliance and ventilation effectiveness in ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed Amyotrophic Lateral Sclerosis (ALS) due to El Escorial criteria
* Must have already established Non-invasive ventilation (NIV)

Exclusion Criteria:

* Ages under 18 years
* Unstable ischemic heart disease
* Oncological disease
* Ventilatory support dependency (more than 16h per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnoea-hypopnea index (AHI) | Baseline, one and three months after the intervention.
  Change in number of apnea and hypopnea events per hour of sleep
Time of NIV use | Baseline, one and three months after the intervention.
  Change in median daily and average daily of hours, minutes
NIV Leaks | Baseline, one and three months after the intervention.
  Change in median and 95%
NIV time of use | Baseline, one and three months after the intervention.
  Change in % of time of use > than 4 hours/day
NIV compliance | Baseline, one and three months after the intervention.
  Change in number of interruptions, complains and ventilator adjustments

SECONDARY OUTCOMES:
Night-time pulseoximeter | Baseline, one and three months after the intervention.
  Change in oxygen saturation of patients blood
Night-time capnography | Baseline, one and three months after the intervention.
  Change in concentration or partial pressure of carbon dioxide in the respiratory gases

CONTACTS AND LOCATIONS:
Overall Officials: Tiina M Andersen, PhD, Principal Investigator — Haukeland University Hospital; Bebiana Conde, PhD fellow, Principal Investigator — Centro Hospitalar Tras-os-Montes e Alto Douro
Locations (2):
- Norwegian National Advisory Unit on Long-term Mechanical Ventilation at Thoracic Department, Haukeland University Hospital, Bergen, Hordaland, Norway
- Centro Hospitalar Tras-os-Montes e Alto Douro, Vila Real, Portugal

IPD SHARING:
Plan to Share IPD: No
Since the study examines patients with a rare disease in the defined geographical areas, we need to be careful not to share data that can be identifiable. A study protocol, informed consent forms and data analysis plan will be available within 6 months of study completion.

REFERENCES:
- [Background] Andersen T, Sandnes A, Brekka AK, Hilland M, Clemm H, Fondenes O, Tysnes OB, Heimdal JH, Halvorsen T, Vollsaeter M, Roksund OD. Laryngeal response patterns influence the efficacy of mechanical assisted cough in amyotrophic lateral sclerosis. Thorax. 2017 Mar;72(3):221-229. doi: 10.1136/thoraxjnl-2015-207555. Epub 2016 May 12. PMID 27174631
- [Background] Andersen TM, Sandnes A, Fondenes O, Nilsen RM, Tysnes OB, Heimdal JH, Clemm HH, Halvorsen T, Vollsaeter M, Roksund OD. Laryngeal Responses to Mechanically Assisted Cough in Progressing Amyotrophic Lateral Sclerosis. Respir Care. 2018 May;63(5):538-549. doi: 10.4187/respcare.05924. Epub 2018 Apr 17. PMID 29666294
- [Background] Andersen TM, Sandnes A, Fondenes O, Clemm H, Halvorsen T, Nilsen RM, Tysnes OB, Heimdal JH, Vollsaeter M, Roksund OD. Laryngoscopy Can Be a Valuable Tool for Unexpected Therapeutic Response in Noninvasive Respiratory Interventions. Respir Care. 2018 Nov;63(11):1459-1461. doi: 10.4187/respcare.06674. No abstract available. PMID 30389835
- [Background] Conde B, Martins N, Brandao M, Pimenta AC, Winck JC. Upper Airway Video Endoscopy: Assessment of the response to positive pressure ventilation and mechanical in-exsufflation. Pulmonology. 2019 Sep-Oct;25(5):299-304. doi: 10.1016/j.pulmoe.2019.02.008. Epub 2019 Apr 16. PMID 31000441
- [Background] Andersen TM, Halvorsen T, Fondenes O, Heimdal JH, Roksund OD, Vollsaeter M, Roksund OD. Larynx: The Complex Gateway to the Lungs. Respir Care. 2019 Jul;64(7):866-869. doi: 10.4187/respcare.06989. No abstract available. PMID 31243162